CLINICAL TRIAL: NCT04352075
Title: Intra Articular Injection of Autologous Microfat and Platelet-rich Plasma in the Treatment of Knee Osteoarthritis: a Pilot Study
Brief Title: Intra Articular Injection of Microfat and PRP in Knee Osteoarthritis
Acronym: MICROPREP
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Clinique Juge (Other)
Responsible Party: Principal Investigator, Marie-Laure LOUIS, Principal investigator, Clinique Juge
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016-004755-75; 2016-004755-75 (EudraCT Number)
Record Dates: First submitted 2020-04-15; First posted 2020-04-17 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Knee Osteoarthritis
Keywords: knee; osteoarthritis; microfat; platelet rich plasma
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Prospective, monocentric randomised, double blind
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Microfat + PRP 3M platelets (Experimental): microfat (5 ml) associated with PRP with a dose of 3 billions of platelets (5 ml)
  Interventions: Drug: Autologous biologic drug of innovative therapy /cell therapy drug
- Microfat + PRP 1M platelets (Experimental): microfat (5 ml) associated with PRP with a dose of 1 billion of platelets (5 ml)
  Interventions: Drug: Autologous biologic drug of innovative therapy /cell therapy drug
- Microfat (Experimental): microfat (5 ml) and saline solution (5 ml)
  Interventions: Drug: Autologous biologic drug of innovative therapy /cell therapy drug

INTERVENTIONS:
Drug: Autologous biologic drug of innovative therapy /cell therapy drug — Articular knee injection of microfat associated with a dose of 3 billions of platelets or associated with a dose of 1 billion of platelets or with saline solution

SUMMARY:
The hypothesis of this project is that the injection of an innovative treatment (microfat and dose of autologous PRP) allows to delay knee arthroplasty in patients with knee OA resistant to medical treatment.

DETAILED DESCRIPTION:
Osteoarthritis is the most common joint disease in the world and one of the most common causes of pain and functional disability. The incidence of cartilage pathology has grown due to the ageing population, and the increase in sports participation and its associated trauma. The treatment of these cartilage damage is limited and remains a major public health issue.

The aim of the medical treatment and intra articular injections consists in reducing pain and improving the knee function in order to limit the sport, professional and social negative impact in the youngest patients. Nevertheless their efficacy remain non predictable in patients.

The arthroplasty will be proposed in the final intention. Insofar arthroplasty is a surgical procedure 1 / which presents a potential infectious risk associated with its invasive nature, 2 / it requires iterative revision surgery, especially in young patients given the limited lifetime of the implants and 3 / whose complete postoperative recovery take several months, it seems justified to continue studies to validate effective alternative treatments to delay the use of joint replacements.

Recently, the emergence of biotherapy in orthopedics has developed the use of intra-articular injections of platelet-rich plasma (PRP). Their use has increased substantially and is based on the demonstration that platelet-rich plasma concentrate growth factors, can stimulate cartilage regeneration in vitro and in vivo preclinical models. In humans, recent data from the literature show that these autologous products are very well tolerated. Their scientific evaluation remains difficult in that 1 / indications and surgical procedures are not harmonized 2 / manufacturing processes PRP are not standardized 3 / quantitative and qualitative composition of PRP is rarely documented.

PRP administration procedures can be optimized: indeed in that, it is a liquid preparation (platelet suspension), its administration in a interface tissue allows to limit its spread and potentiate its trophic effect on the injured cartilage site. Adipose tissue is the most relevant interface tissue given, because it's a tissue rich in stem cells with full therapeutic potential and is easily accessible by subcutaneous minimally invasive procedure. Thus, autologous microfat (fat removed under local anesthesia by manual liposuction using fine cannulas specific) administered in the synovial capsule, could play the matrix to receive the injection of PRP.

The hypothesis of this project is that the standardized injection of an innovative treatment (microfat and dose of autologous PRP) allows to delay knee arthroplasty in patients with knee OA resistant to medical treatment. This treatment, minimally invasive and with economically reasonable cost, would provide a new treatment for second intention. In terms medicoeconomic if this treatment is effective over a period of several years, even in cases where it is necessary to do it one or two times, it would significantly reduce the financial and societal impact of joint replacements.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between 20 to 65 years of age
* Symptomatic knee osteoarthritis , ICRS grade 2, 3 ou 4 with VAS > 4 and failure of medical treatment for at least one year
* BMI between 20 to 30
* Written informed consent, signed by patient or legal representative
* HB > 10g/dl
* Negative pregnancy test
* Social security affiliated

Exclusion Criteria:

* IRM contre-indications: ocular loose bodies, pace maker, neurostimulateur, cochlear implant, vascular clips, mettalic cardiac valve
* BMI < 20
* Thrombocytopenia < 150 G/L
* Thrombocytosis > 450 G/L
* Thrombopathy
* TP < 70%
* TCA patient / witness rapport > 1,20
* Anaemia: HB < 10g/dl
* Positive serology VIH1 and 2, Agp24, Ac HCV, Ag HbS, AcHbc, Ac HTLV I and II, TPHA
* Treatment by platelet inhibiting agent, aspirin, anti vitamin K completed more than 2 weeks before inclusion
* Chronic treatment by corticosteroid per os or treatment completed more than 2 weeks before inclusion
* Intra articular knee injection of corticosteroid more than 8 weeks before inclusion
* Intra articular knee injection of hyaluronic acid more than 8 weeks before inclusion
* NSAI treatment completed more than 2 weeks before inclusion
* Fever or recent disease
* Auto immune disease
* Inflammatory Arthritis
* Immune deficit
* Infectious disease
* Malignant tumor being treated or history of malignant tumor

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Cartilage relaxation time on MRI T2-mapping at 3 months | Baseline and 3 months post injection
  The primary objective of this study is to demonstrate the efficacy of intra-articular injection of autologous microfat associated with a standardized preparation of autologous PRP, by changes in the cartilage relaxation time on MRI T2-mapping at 3 months.

SECONDARY OUTCOMES:
Improved of chondral lesion on MRI | Baseline and 3 and 6 months post injection
  Improved chondral lesions at 3 months and 6 months on specific MRI cartilage sequences (DP FATSAT Axial, Axial T1, T2 mapping): quantitative morphological sequences resolution and qualitative structural sequences.
Pain | Baseline and 1 and 3 and 6 months post injection
  The evolution of pain with the visual analogic scale compared to the initial state (scores at baseline) and the evolution of pain (VAS score) at 1, 3 and 6 months post-injection. Scale from 0 (no pain) to 10 (maximal pain)
Responding patients | Baseline and 3 and 6 months post injection
  The proportion of patients not responding to treatment.
Biologic parameters / clinical efficacity | Baseline and 3 and 6 months post injection
  The correlation between clinical efficacy and dose of PRP administered and dose of growth factors administered.
WOMAC | Baseline and 1 and 3 and 6 months post injection
  The evolution of the functional impact of knee osteoarthritis with the Western Ontario and McMaster University Osteoarthritis score at 1, 3 and 6 months post-injection. Score from 0 to 96 (the worst)

CONTACTS AND LOCATIONS:
Overall Officials: Marie Laure Louis, MD, Principal Investigator — ICOS Corporation
Locations (1):
- Louis, Marseille, France

IPD SHARING:
Plan to Share IPD: No
Publication

REFERENCES:
- [Derived] Louis ML, Dumonceau RG, Jouve E, Cohen M, Djouri R, Richardet N, Jourdan E, Giraudo L, Dumoulin C, Grimaud F, George FD, Veran J, Sabatier F, Magalon J. Intra-Articular Injection of Autologous Microfat and Platelet-Rich Plasma in the Treatment of Knee Osteoarthritis: A Double-Blind Randomized Comparative Study. Arthroscopy. 2021 Oct;37(10):3125-3137.e3. doi: 10.1016/j.arthro.2021.03.074. Epub 2021 Apr 20. PMID 33887408